CLINICAL TRIAL: NCT04525885
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, 12-Month Study to Evaluate the Efficacy and Safety of MK-7264 in Adult Participants With Chronic Cough (PN030)
Brief Title: A Study of Gefapixant (MK-7264) in Adult Participants With Chronic Cough (MK-7264-030)-China Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7264-030 China Extension; MK-7264-030 (Other: Merck Protocol Number); MK-7264-030-02 (Other: Merck Protocol Number)
Record Dates: First submitted 2020-08-18; First posted 2020-08-25 (Actual); Results first posted 2023-10-02 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant; BID protein, human

STUDY DESIGN:
Intervention Model Description: Participants with refractory or unexplained chronic cough will be randomized to 1 of 3 treatment groups: gefapixant 45 mg twice daily (BID), gefapixant 15 mg BID, or placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Gefapixant 45 mg BID (Experimental): Participants will receive a gefapixant 45 mg tablet BID during the main study period (24 weeks) and also during the extension period (28 weeks).
  Interventions: Drug: Gefapixant 45 mg twice daily (BID); Drug: Gefapixant 45 mg BID
- Gefapixant 15 mg BID (Experimental): Participants will receive a gefapixant 15 mg tablet BID during the main study period (24 weeks) and also during the extension period (28 weeks).
  Interventions: Drug: Gefapixant 15 mg BID
- Placebo (Placebo Comparator): Participants will receive a matching placebo tablet BID during the 24-week main study period and during the 28-week extension period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant 45 mg twice daily (BID) — Gefapixant 45 mg tablet to be administered orally BID
  Other Names: MK-7264
  Arms: Gefapixant 45 mg BID
Drug: Gefapixant 15 mg BID — Gefapixant 15 mg tablet to be administered orally BID
  Other Names: MK-7264
  Arms: Gefapixant 15 mg BID
Drug: Placebo — Placebo tablet administered orally BID
  Arms: Placebo
Drug: Gefapixant 45 mg BID — Gefapixant 45 mg tablet to be administered orally BID
  Other Names: MK-7264
  Arms: Gefapixant 45 mg BID

SUMMARY:
The primary objective of this study will be to evaluate the efficacy of gefapixant (MK-7264) in reducing cough frequency as measured over a 24-hour period. It is hypothesized that at least one dose of gefapixant is superior to placebo in reducing coughs per hour (over 24 hours) at Week 24.

DETAILED DESCRIPTION:
This study will have a main 24-week treatment period and a 28-week extension period of treatment. Participants at selected sites and countries who complete the main and extension study periods may consent to participate in an observational, 3-month, Off-treatment Durability Study Period.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiograph or computed tomography scan of the thorax (within 5 years of Screening/Visit 1 and after the onset of chronic cough) not demonstrating any abnormality considered to be significantly contributing to the chronic cough or any other clinically significant lung disease in the opinion of the principal investigator or the sub-investigator
* Has had chronic cough for at least 1 year with a diagnosis of refractory chronic cough or unexplained chronic cough
* Is a female who is not pregnant, not breastfeeding, not of childbearing potential, or agrees to follow contraceptive guidance
* Provides written informed consent and is willing and able to comply with the study protocol (including use of the digital cough recording device and completion of study questionnaires)

Exclusion Criteria:

* Is a current smoker or has given up smoking within 12 months of Screening, or is a former smoker with greater than 20 pack-years
* Has a history of respiratory tract infection or recent clinically significant change in pulmonary status
* Has a history of chronic bronchitis
* Is currently taking an angiotensin converting enzyme inhibitor (ACEI), or has used an ACEI within 3 months of Screening
* Has an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m^2 at Screening OR an eGFR ≥30 mL/min/1.73 m^2 and <50 mL/min/1.73 m^2 at Screening with unstable renal function
* Has a history of malignancy <=5 years
* Is a user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence
* Has a history of anaphylaxis or cutaneous adverse drug reaction (with or without systemic symptoms) to sulfonamide antibiotics or other sulfonamide-containing drugs
* Has a known allergy/sensitivity or contraindication to gefapixant
* Has donated or lost >=1 unit of blood within 8 weeks prior to the first dose of gefapixant
* Has previously received gefapixant or is currently participating in or has participated in an interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (8):
- China (8):
  - The First Affiliated Hospital of Fujian Medical University ( Site 5017), Fuzhou, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 5000), Guangzhou, Guangdong
  - Inner Mongolia Autonomous Region Hospital ( Site 5018), Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Nanchang University ( Site 5012), Nanchang, Jiangxi
  - ShengJing Hospital of China Medical University ( Site 5024), Shenyang, Liaoning
  - Shanghai General Hospital ( Site 5010), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Zhejiang University ( Site 5014), Hangzhou, Zhejiang
  - Peking University Third Hospital ( Site 5005), Beijing

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The China extension study enrolled 161 participants. Of the 161 total participants, 4 were previously enrolled in the global study for MK-7264-030 (NCT03449147). Randomization to the gefapixant 15 mg twice daily (BID) was discontinued during the China enrollment period per protocol amendment 5.
Groups:
- Placebo: Participants received dose-matched placebo tablets twice daily (BID) during the 24-week main study period and 28-week extension period.
- Gefapixant 15 mg BID: Participants received a gefapixant 15 mg tablet BID during the main study period (24 weeks) and also during the extension period (28 weeks). This arm was not included in protocol amendment 5 or later.
- Gefapixant 45 mg Twice Daily (BID): Participants received a gefapixant 45 mg tablet BID during the 24-week main study period and 28-week extension period.
Period: Overall Study
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg Twice Daily (BID)
Started | 68 | 27 | 66
Number Treated | 67 | 27 | 66
Completed | 52 | 21 | 45
Not Completed | 16 | 6 | 21
Not completed — Screen Failure | 1 | 0 | 0
Not completed — Withdrawal by Subject | 14 | 6 | 20
Not completed — Physician Decision | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg Twice Daily (BID) | Total
Number analyzed (Participants) | 67 | 27 | 66 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (15.1) | 44.8 (12.7) | 48.0 (14.5) | 45.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 11 | 32 | 75
  Male | 35 | 16 | 34 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 67 | 27 | 66 | 160
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 67 | 27 | 66 | 160
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline 24-Hour Coughs Per Hour [Mean (Standard Deviation); unit: Coughs/hour] — 24-hour coughs per hour is defined as the average hourly cough frequency based on 24-hour sound recordings using a digital recording device (cough monitor). Population: All participants with 24-hour coughs per hour data available at baseline
  Coughs/hour
    number analyzed (Participants) | 65 | 27 | 65 | 157
    (all) | 29.65 (53.24) | 40.28 (66.66) | 38.62 (49.33) | 35.19 (54.08)

OUTCOME MEASURES:

1. Primary Outcome: Model-Based Geometric Mean Ratio (GMR) of 24-Hour Coughs Per Hour at Week 24
Description: 24-hour coughs per hour was defined as the average hourly cough frequency based on 24-hour sound recordings using a digital recording device (cough monitor). A longitudinal analysis of covariance (ANCOVA) model was applied to log-transformed cough data to determine geometric mean (GM) 24-hour coughs per hour at baseline and week 24. The GMR (Week 24 GM 24-hour coughs per hour divided by Baseline GM 24-hour coughs per hour) is reported.
Time Frame: Baseline, Week 24
Population: All China participants randomized to the gefapixant 45 mg BID or placebo groups who received at least 1 dose of study intervention. Participants needed to have baseline and at least 1 post-baseline measurement. Efficacy evaluation of the gefapixant 15 mg BID group was removed from the study objectives of the China cohort per protocol amendment 5. Participants were analyzed in the group as randomized.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | Gefapixant 45 mg Twice Daily (BID)
Number analyzed (Participants) | 65 | 64
Ratio | 0.47 [0.35 to 0.64] | 0.51 [0.37 to 0.71]
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg Twice Daily (BID); Test type: Superiority — Comparison based on a longitudinal ANCOVA model that included treatment, visit, treatment-by-visit interaction, gender, log-transformed baseline value, and log-transformed baseline value-by-visit as covariates; p = 0.713, ANCOVA; Estimated Relative Reduction (%) = 8.70, 95% CI 2-sided [-30.51 to 70.03] — Estimated relative reduction (ERR) relative to placebo was calculated by 100 (e**DIFF -1), where e**DIFF=exponent of difference; and DIFF= treatment difference in change from baseline at Week 24 based on log transformed data

2. Primary Outcome: Percentage of Participants Who Experienced At Least One Adverse Event (AE) During Treatment and Follow-up
Description: Assessment of participants who have at least one AE during the main study period (24 weeks), the treatment extension period (28 weeks), and during 2 weeks of follow-up by telephone.
Time Frame: Up to 54 weeks
Population: All randomized China participants who received at least 1 dose of study intervention. Participants were analyzed in the group as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg Twice Daily (BID)
Number analyzed (Participants) | 67 | 27 | 66
Participants | 54 | 20 | 58

3. Primary Outcome: Percentage of Participants Who Discontinued Treatment Due to an AE
Description: Assessment of participants who stop study treatment due to an AE during the main study period (24 weeks) or the treatment extension period (28 weeks).
Time Frame: Up 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Gefapixant 45 mg Twice Daily (BID) | Gefapixant 15 mg BID | Placebo
Number analyzed (Participants) | 67 | 27 | 66
Participants | 0 | 1 | 5

4. Secondary Outcome: Model-Based GMR of Awake Coughs Per Hour at Week 24/Baseline
Description: Awake coughs per hour was defined as the average hourly cough frequency while the participant is awake, based on a 24-hour interval of sound recordings using a digital recording device (cough monitor). ANCOVA model was applied to log-transformed cough data to determine GM of awake coughs per hour at baseline and week 24. The GMR (Week 24 GM awake coughs per hour divided by Baseline GM awake coughs per hour) is reported.
Time Frame: Baseline, Week 24
Population: All China participants randomized to the gefapixant 45 mg BID or placebo groups who received at least 1 dose of study intervention. Efficacy evaluation of the gefapixant 15 mg BID group was removed from the study objectives of the China cohort per protocol amendment 5. Participants needed to have awake 24-hour cough data at baseline and at least 1 post-baseline measurement. Participants were analyzed in the group as randomized.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | Gefapixant 45 mg Twice Daily (BID)
Number analyzed (Participants) | 65 | 64
Ratio | 0.46 [0.33 to 0.62] | 0.51 [0.37 to 0.70]
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg Twice Daily (BID); Test type: Superiority; p = 0.628, ANCOVA — Comparison based on a longitudinal ANCOVA model that included treatment, visit, treatment-by-visit interaction, gender, log-transformed baseline value, and log-transformed baseline value-by-visit as covariates; Estimated Relative Reduction (%) = 11.58, 95% CI 2-sided [-28.68 to 74.57] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With a ≥1.3-point Increase From Baseline in the Leicester Questionnaire (LCQ) Total Score at Week 24
Description: The 19-item LCQ assessed the impact of chronic cough in three health-related quality of life (HRQoL) domains (physical, social and psychological). The LCQ is calculated as a mean score for each domain ranging from 1 to 7, with a total score ranging from 3 to 21. Higher scores indicate better HRQoL. A clinically meaningful improvement from baseline in HRQoL was defined as ≥1.3-point increase in the LCQ total score at Week 24. The percentage of participants (logistic regression model-based) with a ≥1.3-point increase in the LCQ total score at Week 24 is presented.
Time Frame: Baseline, Week 24
Population: All China participants randomized to the gefapixant 45 mg BID or placebo groups who received at least 1 dose of study intervention. Efficacy evaluation of the gefapixant 15 mg BID group was removed from the study objectives of the China cohort per protocol amendment 5. Participants needed to have LCQ data at baseline and at least 1 post-baseline measurement. Participants were analyzed in the group as randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 45 mg Twice Daily (BID)
Number analyzed (Participants) | 67 | 64
Percentage of Participants | 68.4 | 67.5
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg Twice Daily (BID); Test type: Superiority; p = 0.917, Regression, Logistic — Comparison based on logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, baseline LCQ total score, and the interaction of baseline LCQ total score by visit as covariates; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.43 to 2.13]

6. Secondary Outcome: Percentage of Participants With a ≥30% Reduction From Baseline in 24-hour Coughs Per Hour at Week 24
Description: 24-hour coughs per hour was defined as the average hourly cough frequency based on 24-hour sound recordings using a digital recording device (cough monitor). A clinically meaningful improvement from baseline is defined as a ≥30% reduction in 24-hour coughs per hour at week 24. The percentage of participants (logistic regression model-based) with a ≥30% reduction from baseline in 24-hour coughs per hour at Week 24 (≥30% reduction from baseline) is presented.
Time Frame: Baseline, Week 24
Population: All China participants randomized to the gefapixant 45 mg BID or placebo groups who received at least 1 dose of study intervention. Efficacy evaluation of the gefapixant 15 mg BID group was removed from the study objectives of the China cohort per protocol amendment 5. Participants needed to have 24-hour cough data at baseline and at least 1 post-baseline measurement. Participants were analyzed in the group as randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 45 mg Twice Daily (BID)
Number analyzed (Participants) | 65 | 64
Percentage of Participants | 54.6 | 50.6
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg Twice Daily (BID); Test type: Superiority; p = 0.687, Regression, Logistic — Comparison based on a logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, baseline 24-hour coughs per hour and the interaction of baseline 24-hour coughs per hour by visit as covariates; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.38 to 1.88]

7. Secondary Outcome: Percentage of Participants With ≥1.3-point Reduction From Baseline of Mean Weekly Cough Severity Diary (CSD) Total Score at Week 24
Description: The 7-item CSD was used to record participants' daily cough frequency, cough intensity, and disruption due to cough. Each item was rated on an 11-point scale ranging from 0 (best) to 10 (worst); the total daily CSD score was the sum of these seven item scores (Min=0, Max=70). Mean weekly CSD total score was defined as the average of the mean total daily scores collected during the week prior to each visit. The percentage of participants (logistic regression model-based) with a ≥1.3 point reduction from baseline in CSD at Week 24 is reported.
Time Frame: Baseline, Week 24
Population: All China participants randomized to the gefapixant 45 mg BID or placebo groups who received at least 1 dose of study intervention. Efficacy evaluation of the gefapixant 15 mg BID group was removed from the study objectives of the China cohort per protocol amendment 5. Participants needed to have CSD data at baseline and at least 1 post-baseline measurement. Participants were analyzed in the group as randomized.
Measure: Number; unit: Percentage of Participants
Groups:
- Gefapixant 45 mg BID: Participants received a gefapixant 45 mg tablet BID during the 24-week main study period and 28-week extension period.
Arm/Group | Placebo | Gefapixant 45 mg BID
Number analyzed (Participants) | 65 | 62
Percentage of Participants | 58.7 | 61.1
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg BID; Comparison based on a logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, baseline mean weekly CSD total score and the interaction of baseline mean weekly CSD total score by visit as covariates; Test type: Other; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.49 to 2.49]

8. Secondary Outcome: Percentage of Participants With ≥2.7-point Reduction From Baseline of Mean Weekly CSD Total Score at Week 24
Description: The 7-item CSD was used to record participants' daily cough frequency, cough intensity, and disruption due to cough. Each item was rated on an 11-point scale ranging from 0 (best) to 10 (worst); the total daily CSD score was the sum of these seven item scores (Min=0, Max=70). Mean weekly CSD total score was defined as the average of the mean total daily scores collected during the week prior to each visit. The percentage of participants (logistic regression model-based) with a ≥2.7 point reduction from baseline in CSD at Week 24 is reported.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 45 mg BID
Number analyzed (Participants) | 65 | 62
Percentage of Participants | 23.9 | 37.8
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg BID; Comparison based on a logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, baseline mean weekly CSD total score, and the interaction of baseline mean weekly CSD total score by visit as covariates; Test type: Other; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.80 to 4.64]

9. Secondary Outcome: Percentage of Participants With a ≥30 mm Reduction From Baseline in Cough Severity Visual Analog Scale (VAS) Score at Week 24
Description: The VAS is a single-item questionnaire with the response on a 100- point scale ranging from 0 ("No Cough") to 100 ("Extremely Severe Cough"). Mean weekly VAS score was defined as the average of the VAS scores collected during the week prior to each visit. The percentage of participants (logistic regression model-based) with a ≥30mm reduction from baseline in cough severity VAS score at Week 24 is reported.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Groups:
- Gefapixant 45 BID: Participants received a gefapixant 45 mg tablet BID during the 24-week main study period and 28-week extension period.
Arm/Group | Placebo | Gefapixant 45 BID
Number analyzed (Participants) | 65 | 62
Percentage of Participants | 23.0 | 24.9
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 BID; Test type: Other — Comparison based on a logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, baseline mean weekly VAS score, and the interaction of baseline mean weekly VAS score by visit as covariates; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.45 to 2.72]

ADVERSE EVENTS:
Time Frame: Up to approximately 54 weeks
Description: All-cause mortality (ACM) population includes all randomized participants; Serious and other AEs include all randomized participants who took ≥1 one dose of study drug.
Groups:
- MK-7264 15 mg BID: Participants received a gefapixant 15 mg tablet and placebo tablet to match gefapixant 45 mg BID during the 24-week main study period and 28-week extension period.
- MK-7264 45 mg BID: Participants received a gefapixant 45 mg tablet and placebo tablet to match gefapixant 15 mg BID during the 24-week main study period and 28-week extension period.
Arm/Group | Placebo | MK-7264 15 mg BID | MK-7264 45 mg BID
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/27 | 0/66
Serious Adverse Events (participants affected / at risk) | 4/67 | 4/27 | 2/66
Other Adverse Events (participants affected / at risk) | 42/67 | 17/27 | 53/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=67) | MK-7264 15 mg BID (N=27) | MK-7264 45 mg BID (N=66)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis gastrointestinal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=67) | MK-7264 15 mg BID (N=27) | MK-7264 45 mg BID (N=66)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 4 (5) | 2 (3)
Chest pain (General disorders) | 5 (7) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (5) | 3 (5) | 3 (4)
Nasopharyngitis (Infections and infestations) | 3 (4) | 2 (4) | 3 (5)
Pharyngitis (Infections and infestations) | 7 (7) | 1 (1) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 14 (23) | 4 (5) | 10 (11)
Accidental overdose (Injury, poisoning and procedural complications) | 5 (8) | 2 (2) | 5 (6)
Crystal urine (Investigations) | 6 (7) | 0 (0) | 4 (4)
Crystal urine present (Investigations) | 7 (7) | 2 (3) | 7 (9)
Urinary occult blood positive (Investigations) | 2 (2) | 2 (2) | 2 (2)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 6 (6)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 12 (12)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Haematuria (Renal and urinary disorders) | 8 (10) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3) | 11 (12)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship should reflect significant contribution to the design and conduct of the trial, performance or interpretation of the analysis, and/or writing of the manuscript. All named authors must be able to defend the trial results and conclusions. MSD funding of a trial will be acknowledged in publications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT04525885/Prot_SAP_000.pdf